CLINICAL TRIAL: NCT01131702
Title: Randomized,2-way Crossover, Bioequivalence Study of Ranitidine 300 mg Tablets Zantac 300 mg Tablets Administered as 1 x 300 mg Tablet in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalency Study of Ranitidine Tablets 300 mg of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Dr. Ramakrishna Bangaru/Assistant Manager, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 02399
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Ranitidine
MeSH Terms: interventions — Ranitidine; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranitidine Tablets, 300 mg (Experimental): Ranitidine Tablets, 300 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Ranitidine
- Zantac Tablets, 300 mg (Active Comparator)
  Interventions: Drug: Ranitidine

INTERVENTIONS:
Drug: Ranitidine — Ranitidine Tablets, 300 mg
  Other Names: Zantac 300 mg tablets of Glaxosmithkline

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of ranitidine 300 mg tablets versus Zantac 300 mg tablets administered as 1 x 300 mg tablet under fasting conditions.

DETAILED DESCRIPTION:
This study compared the rate and extent of absorption of ranitidine 300 rng tablets versus Zantac. The study products were administered as a single oral dose of 1 x 300 mg tablet using a randomized, two-way crossover fasting study in non-smoker healthy volunteers with a washout period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may be done using different media (e.g. radio, newspaper, Anapharm Inc. Web site. Anapharm Inc. volunteers' data base). Subjects must meet all of the following criteria in order to be included in the study:

  * Subjects will be females and/or males, non-smokers, 18 years of age and older.

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  * Clinically significant illnesses within 4 weeks of the administration of study medication.
  * Clinically significant surgery within 4 weeks prior to the administration of the study medication.
  * Any clinically significant abnormality found during medical screening.
  * Any reason which, in the opinion of the medical sub investigator would prevent the subject from participating in the study.
  * Abnormal laboratory tests judged clinically significant.
  * Positive urine drug screen at screening.
  * Positive testing for hepatitis B, hepatitis C or HIV at screening.
  * ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90 mmHg; or heart rate less than 50 or over 100 bpm) at screening.
  * Subjects with BMI ≥ 30.0.
  * History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
  * History of-drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
  * History of allergic reactions to ranitidine or other Hr receptor antagonists (e.g.cimetidine, famotidine, nizatidine).
  * History of allergic reactions to heparin.
  * Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates. carbamazepine. phenytoin. glucocorticoids rifampin/rifabutin;examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin ketoconazole, MAO inhibitors, neuroleptics, verapamil. quinidine) within 30 days prior to administration of the study medication.
  * Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
  * History or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea inflammatory bowel diseases)unresolved gastrointestinal symptoms (e.g.diarrhea, vomiting), liver or kidney disease or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
  * Any history or presence of clinically significant neurological, endocrinal, cardiovascular,pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
  * Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
  * Use of any tobacco products in the last 6 months.
  * Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical sub investigator, contraindicates the subject's participation in this study.
  * Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
  * Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows:
  * less than 300 niL of whole blood within 30 days or
  * 300 mL to 500 mL of whole blood within 45 days or
  * more than 500 mL of whole blood within 56 days.
  * Subjects with history or known presence of porphyria.

Additional exclusion criteria for females only:

* Breast-feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).
* Female subjects of childbearing potential who have had unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. The acceptable methods of contraception are:

  * Condom + spermicide
  * Diaphragm +spermicide
  * Intrauterine contraceptive device (placed at least 4 weeks prior to study drug administration).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-01; Primary Completion 2003-02 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bicrell, M.D., Principal Investigator — Anapbarm Inc.
Locations (1):
- Anapharm Inc., Montreal, Quebec, Canada